CLINICAL TRIAL: NCT04743284
Title: The Agreement Between Face-to-Face and Tele-Assessment of Balance Tests in Patient With Multiple Sclerosis
Brief Title: Tele-Assessment and Face-to-Face Evaluation of Balance in MS
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst. Prof., Istanbul University - Cerrahpasa
Other Study IDs: E-71938118-604.01.01-52315
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: Tele-medicine; Neurorehabilitation; Stability; Gait; Questionnaire
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tele-assessment: The balance evaluations will be applied by the tele-assessment method.
- face-to-face assessment: The balance evaluations will be applied by the face-to-face assessment method in a clinical setting

SUMMARY:
MS is characterized by clinical symptoms caused by lesions of the brain, spinal cord, or optic nerves that can affect balance, gait, and risk of falls. 50-80% of patients with MS have different levels of balance-related pathological findings. In addition, the imbalance is one of the most complained about findings by MS patients.

Balance and postural control disorders are the most common signs in patients with cerebellar tract damage. Many patients have reported problems with balance and gait causing serious disability. Therefore, disorders of balance and postural control in patients with MS are associated with difficulty in standing and performing functional activities. Effective quantitative methods are needed to assess postural imbalance to help clinicians assess the progression of this disorder.

Current literature suggests that home tele-rehabilitation and tele-medicine practices may be an alternative method effective enough to be equivalent to face-to-face physiotherapy treatments for patients with Ms. The advantages of Tele-medicine over normal care include increased social support, participant engagement, quality of care, cost-effectiveness, access to services (due to lack of transportation), and reducing the burden on healthcare professionals to make services easier to deploy. In cases such as Pandemic conditions, where face-to-face service is disrupted in clinics, tele-rehabilitation can be applied as a suitable alternative treatment method accessible to patients. The effectiveness of Tele-rehabilitation raises the question of whether tele-evaluation is as effective and accurate as in the clinic. Studies examining the effectiveness of Tele-assesment are still insufficient. The study is planned to address this deficiency.

The aim of this study is to compare the results of MS patients by applying valid and reliable methods used in balance assessment with face-to-face and online access methods, thereby investigating the effectiveness of balance assessment through online access.

The hypothesis in this study is that the results of the balance assessment with online access in MS patients will be consistent with the results of the balance assessment conducted face-to-face.

H0: Tele-assessments of balance do not give the same results as face-to-face balance assessments in MS patients.

H1: Tele-assessments of balance do not give the same results as face-to-face balance assessments in MS patients.

DETAILED DESCRIPTION:
Voluntary patients who have been diagnosed with MS will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. Tele-assessment will be applied to one group first, and face-to-face assessment will be applied to the other group first.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Patients diagnosed with MS according to McDonald diagnostic criteria with an EDSS score of 0-6
* Internet presence in the environment where they will perform the evaluation
* Having an internet-based technological tool or having access to this tool
* Having someone to accompany the patient during the evaluation
* Agree to participate in the study
* Ability to understand and speak Turkish

Exclusion Criteria:

* Having had a new attack in the last 3 months
* Use high-dose corticosteroid therapy in the last 2 weeks
* Presence of orthopedic problems/problems that can cause balance problems
* Having cognitive disorders that will prevent him from communicating
* Having a level of visual and auditory problems that will prevent communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with MS
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | change from baseline at 3rd day
  It is a scale containing 14 instructions and a score of 0-4 is given by observing the patient's performance for each instruction. 0 points are given in cases where the patient cannot perform the activity at all, while 4 points are given when the patient completes the activity independently. The highest score is 56 and 0-20 points indicate balance disorder, 21-40 points indicate an acceptable balance, 41-56 points indicate the presence of a good balance. It takes between 10 and 20 minutes to complete the scale.
Dynamic Gait Index | change from baseline at 3rd day
  The scale measures mobility function and dynamic balance. The eight tasks of this scale include walking, walking with head turns, turning, walking over objects, walking around objects, and climbing up stairs. The performance is rated on a 4-point scale.
Timed Up and Go Test | change from baseline at 3rd day
  The test is a measure of dynamic balance. It requires individuals to get up from a chair, walk 3 feet, turn and sit. The time from the moment the individual lifts the pelvis from the chair until he or she returns with the pelvis in the chair is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Asst.Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Korn T. Pathophysiology of multiple sclerosis. J Neurol. 2008 Dec;255 Suppl 6:2-6. doi: 10.1007/s00415-008-6001-2. PMID 19300953
- [Background] Browne P, Chandraratna D, Angood C, Tremlett H, Baker C, Taylor BV, Thompson AJ. Atlas of Multiple Sclerosis 2013: A growing global problem with widespread inequity. Neurology. 2014 Sep 9;83(11):1022-4. doi: 10.1212/WNL.0000000000000768. No abstract available. PMID 25200713
- [Background] Mazumder R, Murchison C, Bourdette D, Cameron M. Falls in people with multiple sclerosis compared with falls in healthy controls. PLoS One. 2014 Sep 25;9(9):e107620. doi: 10.1371/journal.pone.0107620. eCollection 2014. PMID 25254633
- [Background] Cameron MH, Nilsagard Y. Balance, gait, and falls in multiple sclerosis. Handb Clin Neurol. 2018;159:237-250. doi: 10.1016/B978-0-444-63916-5.00015-X. PMID 30482317
- [Background] Ilg W, Synofzik M, Brotz D, Burkard S, Giese MA, Schols L. Intensive coordinative training improves motor performance in degenerative cerebellar disease. Neurology. 2009 Dec 1;73(22):1823-30. doi: 10.1212/WNL.0b013e3181c33adf. Epub 2009 Oct 28. PMID 19864636
- [Background] Nelson SR, Di Fabio RP, Anderson JH. Vestibular and sensory interaction deficits assessed by dynamic platform posturography in patients with multiple sclerosis. Ann Otol Rhinol Laryngol. 1995 Jan;104(1):62-8. doi: 10.1177/000348949510400110. PMID 7832544
- [Background] Amatya B, Galea MP, Kesselring J, Khan F. Effectiveness of telerehabilitation interventions in persons with multiple sclerosis: A systematic review. Mult Scler Relat Disord. 2015 Jul;4(4):358-69. doi: 10.1016/j.msard.2015.06.011. Epub 2015 Jun 19. PMID 26195057
- [Background] Bove R, Garcha P, Bevan CJ, Crabtree-Hartman E, Green AJ, Gelfand JM. Clinic to in-home telemedicine reduces barriers to care for patients with MS or other neuroimmunologic conditions. Neurol Neuroimmunol Neuroinflamm. 2018 Oct 2;5(6):e505. doi: 10.1212/NXI.0000000000000505. eCollection 2018 Nov. PMID 30775409
- [Background] Jennett PA, Affleck Hall L, Hailey D, Ohinmaa A, Anderson C, Thomas R, Young B, Lorenzetti D, Scott RE. The socio-economic impact of telehealth: a systematic review. J Telemed Telecare. 2003;9(6):311-20. doi: 10.1258/135763303771005207. PMID 14680514
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Lord SE, Wade DT, Halligan PW. A comparison of two physiotherapy treatment approaches to improve walking in multiple sclerosis: a pilot randomized controlled study. Clin Rehabil. 1998 Dec;12(6):477-86. doi: 10.1191/026921598675863454. PMID 9869251
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Cattaneo D, Jonsdottir J, Repetti S. Reliability of four scales on balance disorders in persons with multiple sclerosis. Disabil Rehabil. 2007 Dec 30;29(24):1920-5. doi: 10.1080/09638280701191859. Epub 2007 Apr 26. PMID 17852286
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576